CLINICAL TRIAL: NCT01011192
Title: Performance of Two Different Ke0s in the Same Pharmacokinetic Propofol Model. Study on Loss and Recovery of Consciousness
Brief Title: Performance of Two Different ke0s in the Same Pharmacokinetic Propofol Model
Status: Completed | Type: Observational
Sponsor: Centro Medico Campinas (Other)
Collaborators: Hospital Santa Sofia Ltda (Unknown)
Responsible Party: Eduardo Tadeu Moraes Santos, Hospital Santa Sofia Ltda
Other Study IDs: RFS 02
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Unconsciousness
Keywords: Intravenous anesthesia; propofol; pharmacokinetic model; Monitoring; bispectral index.
MeSH Terms: conditions — Unconsciousness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ke0 of 0.26 min-1: Individual volunteers using Marsh's pharmacokinetic target-controlled infusion model with ke0 of 0.26 min-1 (Asena PK® - Cardinal Health)
- ke0 of 1.21 min-1: Individual volunteers using Marsh's pharmacokinetic target-controlled infusion model with ke0 of 1.21 min-1 (Primea Orchestra® - Fresenius-Kabi basis)

SUMMARY:
The aim of this study was to assess the clinical performance of two different ke0s (fast and slow) in terms of propofol effect-site concentration (Ce) during the loss and recovery of consciousness, using Marsh's pharmacokinetic model.The hypothesis to be tested was that the Ce of propofol predicted by the slow ke0 in the loss and recovery of consciousness is similar, differently from the fast ke0.

DETAILED DESCRIPTION:
Introduction: The ke0 can be defined as the proportional variation of the gradient of concentration between the plasma and the effect-site in relation to the unit of time. Theoretically, the higher the value of the ke0, the faster the drug enters the effect-site. Therefore, drugs with short T½ke0 have high ke0s and fast onset of action. The aim of this study was to assess the clinical performance of two different ke0s (fast and slow) in terms of propofol effect-site concentration (Ce) during the loss and recovery of consciousness, using Marsh's pharmacokinetic model. Method: Twenty healthy male adult volunteers participated in this study. Propofol was first administered to the individual volunteer using Marsh's pharmacokinetic target-controlled infusion model with ke0 of 1.21 min-1 and, on another opportunity, with the same pharmacokinetic model but ke0 of 0.26 min-1. Propofol was infused in plasma target-concentration of 3.0 µg.mL-1. Loss and recovery of consciousness was defined as response of the volunteer to verbal stimulus. The Ce was registered at the moments of loss and recovery of consciousness. Results: At loss and recovery of consciousness, propofol Ce means predicted by the fast ke0 were different (3.64 ± 0.78 and 1.47 ± 0.29 µg.mL-1, respectively, p < 0.0001), whereas with the slow ke0 the predicted Ce means were similar (2.20 ± 0.70 and 2.13 ± 0.43 µg.mL-1, respectively, p = 0.5425). Conclusion: It can be concluded that slow ke0 (0.26 min-1) incorporated into Marsh's pharmacokinetic model showed better clinical performance than fast ke0 (1.21 min-1), since the predicted effect-site concentrations of propofol at loss and recovery of consciousness were similar.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* male
* adult between 20 and 45 years old

Exclusion Criteria:

* use of alcohol or illicit drugs
* chronic use of H2 inhibitors and tricyclic antidepressants of calcium channel blockers
* hypersensitivity to the drugs used in the experimental protocol.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty healthy male adult volunteers participated in this study. The volunteers appeared at the testing location, having refrained from eating and drinking for six hours. All the volunteers were monitored with electrocardiogram (DII and V1 derivation), pulse oximetry (SpO2), non-invasive average arterial pressure and bispectral index (BIS). Oxygen under 2.0 L.min-1 nasal catheter was used and the left antecubital vein was punctured and connected to the venous catheter filled with propofol (Propovan® - Cristália Laboratório Ltda).
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Propofol effect-site concentration (Ce) during the loss and recovery of consciousness with fast and slow keo. | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Simoni, MD, Principal Investigator — Centro Medico Campinas
Locations (1):
- Hospital Santa Sofia, Campinas, São Paulo, Brazil

REFERENCES:
- [Result] Iwakiri H, Nishihara N, Nagata O, Matsukawa T, Ozaki M, Sessler DI. Individual effect-site concentrations of propofol are similar at loss of consciousness and at awakening. Anesth Analg. 2005 Jan;100(1):107-110. doi: 10.1213/01.ANE.0000139358.15909.EA. PMID 15616062